CLINICAL TRIAL: NCT01192243
Title: Phase 2 Study of Gefitinib Compared With Pemetrexed/Cisplatin in Advanced Non-Small
Brief Title: Study of Gefitinib Compared With Pemetrexed/Cisplatin in Advanced Non-Small Cell Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University Cancer Hospital, Department of Medical Oncology,Fudan University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Iressa combined with Pem/Cis
Record Dates: First submitted 2010-08-04; First posted 2010-09-01 (Estimated); Last update posted 2010-09-03 (Estimated); Status verified 2010-09

CONDITIONS: Toxicity; Non-small Cell Lung Cancer
Keywords: Objective response rate; Time to Progression; Quality of Live
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gefitinib — 250mg qd po d3-16
Drug: Pemetrexed — 500mg/m2 venous infusion,D1,q3w
Drug: Cisplatin or carboplatin — Cisplatin:75mg/m2, venous infusion,D1,q3w or Carboplatin: AUC 5, venous infusion, D1,q3w

SUMMARY:
The purpose of this study is to examine the efficacy and safety of gefitinib combinated with Pemetrexed/Cisplatin in advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed by the histologic, cytologic diagnosis of IV non-small cell lung cancer
* Age from 18 to 70 years old
* At least one target lesion diameter spiral CT ≥ 1 cm, or the common CT ≥ 2 cm, and can be measured by imaging tools
* ECOG 0-1
* Expected life time longer than 12 weeks
* Normal laboratory values:

leucocyte≥ 4×109/L neutrophil≥ 1.5×109/L platelet≥100×109/L Hemoglobin≥ 10g/L ALT and AST ≤2.5×ULN (≤5×ULN if liver metastasis)

Exclusion Criteria:

* Patients have not used drugs according to protocol
* Patients were allergic to pemetrexed or cisplatin
* Patients received radiotherapy or other biological treatment 4 weeks before the trial
* Uncontrolled hydrothorax or hydropericardium
* neuropathy toxicity ≥ CTC 3
* Severe symptomatic heart disease
* Active upper gastrointestinal ulcer or digestive disfunction
* Severe infection or metabolic disfunction
* Patients with other malignant tumor
* Uncontrolled brain metastases
* Patients have accepted other clinical trials
* Female patients during their pregnant and lactation period, or patients without contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
response rate | six weeks

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | six weeks
  according to NCI CTC V3.0
Progression free survival | six weeks
quality of life | six weeks
  according to FACT-LCS scores

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Chang, MD,PhD, Principal Investigator — Fudan University affiliated cancer hospital
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China